CLINICAL TRIAL: NCT05918393
Title: A Behavioral Economic Approach to Improving Communication Variability and Treatment Efficacy
Brief Title: Behavioral Economics and Communication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 941605-12
Record Dates: First submitted 2023-06-02; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Problem Behavior
MeSH Terms: conditions — Problem Behavior

STUDY DESIGN:
Intervention Model Description: Single-case research design including multielement and reversal strategies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functional communication training (FCT) (Other): During FCT, signaled intervals of reinforcement (i.e., the functional reinforcer is available contingent on communication) and extinction (i.e., the functional reinforcer is unavailable and thus both severe destructive behavior (SDB) and communication are on extinction) will be alternated within a single session. During the treatment-challenge evaluation, SDB will remain on extinction throughout and all communication responses will be reinforced on an FR-1 schedule during the signaled reinforcement intervals.
  Interventions: Behavioral: functional communication training

INTERVENTIONS:
Behavioral: functional communication training — During functional communication training, signaled intervals of reinforcement (i.e., the functional reinforcer is available contingent on communication) and extinction (i.e., the functional reinforcer is unavailable and thus both problem behavior and communication are on extinction) will be alternated within a single session. All communication responses will be reinforced every time they occur during the signaled reinforcement intervals.
  Other Names: differential reinforcement

SUMMARY:
This project examines mechanisms to address two significant challenges present in communication-based behavioral interventions for individuals with autism and comorbid severe destructive behavior (SDB): (a) inflexible communication responding and (b) reemergence of severe destructive behavior when challenges to treatment integrity occur. Achieving the proposed aims will advance clinical practice related to the treatment of SDB and generalization of treatment effects to mitigate against the resurgence of SDB

DETAILED DESCRIPTION:
Approximately 25% of individuals with autism spectrum disorder (ASD) are affected by co-morbid severe destructive behavior (SDB). Although there is an extensive body of literature supporting the use of behavioral interventions for decreasing the occurrence of SDB, challenges in the clinical application of these interventions still exist. The current research proposes to evaluate mechanisms for mitigating two potentially significant treatment challenges: (a) invariant responding and (b) resurgence of problem behavior. Functional Communication Training (FCT) is a common reinforcement-based treatment for SBD that involves reinforcement of a target communication response to replace SDB such that communication produces the desired behavior outcome and SDB does not. However, in typical practice only a single communication response is taught thus limiting an individual's ability to communicate if that response is not observed (e.g., touching a card) or if the device used for communication fails (e.g., iPad battery dies). Furthermore, a core deficit of ASD is engagement in restrictive patterns of behavior; thus, individuals with ASD might show a preference for only emitting one communication response among concurrently available alternatives. As noted above, if the preferred communication modality is unavailable, an individual may revert back to engaging in SDB rather than using another, more appropriate communication response - a condition generally referred to as treatment relapse. Evidence for such outcomes can be found in studies in which a FCT response is placed on extinction (i.e., the response no longer produces reinforcement) and SDB immediately increases. One potential way to mitigate against such issues is to teach multiple FCT responses. That is, teaching multiple communication responses may inoculate the individual against invariant communication responding thus reducing SDB.

Related to this, a preferred clinical practice in treating SDB with FCT is to teach the individual to tolerate delays to reinforcement following communication (e.g., waiting until the caregiver is available to interact with the child). When communication is not immediately reinforced, there exists an additional possibility of treatment relapse. Resurgence is one type of treatment relapse in which a previously reduced response re-emerges as a result of a procedural change. For example, relapse of SDB is a clinical concern often observed when delays to reinforcement are introduced. That is, when immediate reinforcement is no longer provided contingent on the target communication response, the individual might revert to engaging in SDB. Given that only one communication response is typically taught during FCT, the effects of teaching multiple communication responses on the mitigation of resurgence remains unknown.

Mitigating invariant responding and resurgence has the potential to greatly impact the lives of individuals with ASD affected by SDB by helping to ensure that positive treatment outcomes maintain across time even in the presence of challenges to treatment such as procedural integrity errors and delays to obtaining reinforcement for appropriate behavior. Thus, the proposed research seeks to strengthen the current literature base and advance current clinical practice through completion of the following aims:

Aim 1. Identify multiple functionally equivalent communication responses and assess levels of variant responding under rich schedule requirements.

Aim 2. Evaluate the effects of a behavioral economic analysis on changes in variant communication responding across multiple communication responses across progressively leaner schedule requirements.

Aim 3. This aim is exploratory in nature as we will assess the extent to which we observe resurgence of SDB following the introduction of multiple communication responses and manipulation of reinforcement schedules for the various responses.

ELIGIBILITY:
Inclusion Criteria:

* between 5 and 13 years of age
* documented diagnosis of autism spectrum disorder (ASD) or a diagnosis confirmed based on the relevant cutoff score of the Autism Diagnostic Observation Scale (ADOS-2)
* referred for clinical assessment and treatment of severe destructive behavior (SDB; e.g., SIB, aggression) that (a) poses a serious danger to self, others, or the environment, and (b) interferes with the child receiving an appropriate education
* children whose functional analysis results indicate that SDB is maintained by social-negative or social-positive reinforcement will be admitted to this investigation.

Exclusion Criteria:

* severity of their SDB prohibits exposure to baseline conditions
* undergoing changes in their medication regimen
* results of the functional analyses indicate that their SDB is maintained by automatic reinforcement

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Appropriate communication | 3-5 days per week for approximately 12 weeks
  Appropriate communication responses for each participant will be selected based on language level as identified via the Peabody Picture Vocabulary Test, 4th edition (PPVT-4) and/or the Expressive Vocabulary Test-3rd edition (EVT-3)
Problem behavior | 3-5 days per week for approximately 12 weeks
  Individualized operational definitions of problem behavior will be developed for each participant. Examples include aggression, disruption, pica, and self-injurious behavior. These data will be determined by clinical interview and measured via direct observation. There are no formal questionnaires, rating scales, or other measures associated with this outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No